CLINICAL TRIAL: NCT00468572
Title: Affectionate Communication as a Mechanism for Responding to Acute Stress
Brief Title: Using Affectionate Communication as a Response to Acute Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Kory Floyd/PI, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: R03MH075757 (NIH); R03MH075757 (NIH); DATR A2-A1A
Record Dates: First submitted 2007-05-01; First posted 2007-05-02 (Estimated); Last update posted 2012-01-10 (Estimated); Status verified 2012-01

CONDITIONS: Stress
Keywords: Emotion; Oxytocin; Cortisol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Participants will receive treatment with affectionate writing
  Interventions: Behavioral: Affectionate Writing
- 2 (Active Comparator): Participants will receive treatment with meaningless writing
  Interventions: Behavioral: Meaningless Writing

INTERVENTIONS:
Behavioral: Affectionate Writing — Participants assigned to the experimental group will spend 20 minutes writing an affectionate letter to a loved one. Levels of cortisol will be measured using saliva samples from each participant during the writing session. Levels of oxytocin, a hormone known to transmit signals within the brain and often associated with bonding and building trusting relationships, will be measured from blood samples taken during the writing session as well.
  Arms: 1
Behavioral: Meaningless Writing — Participants assigned to the control group will spend 20 minutes writing about meaningless topics. Participants will undergo the same testing during the writing session as the experimental group.
  Arms: 2

SUMMARY:
This study will examine the effects of tending to significant social relationships on managing and reducing stress.

DETAILED DESCRIPTION:
Stress is a large part of daily modern life; however, it can cause a number of long-term problems for mental and physical health. Recent research has confirmed that there are definite mental and physical health benefits of maintaining significant positive social bonds. Many of these benefits appear to be associated with the ability to regulate stress that is caused by environmental challenges. Drawing on close relationships and expressing affection may help people to recover from stress more effectively. This study will evaluate the tend-and-befriend theory, which suggests that engaging in behaviors aimed at maintaining and strengthening significant social bonds can act as an adaptive response to acute stress.

All participants in this study will undergo a series of standard laboratory stressors designed to elevate cortisol levels. Cortisol, also known as the "stress hormone," is activated and secreted within the body in response to stress. Current research suggests that displaying signs of affection toward a loved one can lower cortisol levels, causing the body to relax and recover from a stressful situation more quickly. After lab tests have been completed, participants will be randomly assigned to an experimental or control group. Participants assigned to the experimental group will spend 20 minutes writing an affectionate letter to a loved one. Participants assigned to the control group will spend 20 minutes writing about meaningless topics. Levels of cortisol will be measured using saliva samples from each participant during the writing session. Levels of oxytocin, a hormone known to transmit signals within the brain and often associated with bonding and building trusting relationships, will be measured from blood samples taken during the writing session as well. Participants will also provide a self-report of their current stress level at the end of the study. Participation in this study will last approximately 2 hours. By examining associations between the communication of affection and responses to acute stress, this study may eventually lead to the development of new and better treatment options for people with constant acute stress.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Weigh at least 110 pounds
* Moderate to no anxiety about having blood drawn

Exclusion Criteria:

* Hypertension or diabetes
* Current or recent pregnancy
* Colorblindness
* History of cancer
* Current use of alpha blockers, beta blockers, or steroids

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2007-02; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Oxytocin levels | Measured at Hour 2
Cortisol levels | Measured at Hour 2

SECONDARY OUTCOMES:
Self-reported stress level | Measured at Hour 2

CONTACTS AND LOCATIONS:
Overall Officials: Kory Floyd, PhD, Principal Investigator — Arizona State University
Locations (1):
- Exercise and Sports Research Institute, Tempe, Arizona, United States

REFERENCES:
- [Background] Floyd K, Mikkelson AC, Tafoya MA, Farinelli L, La Valley AG, Judd J, Haynes MT, Davis KL, Wilson J. Human affection exchange: XIII. Affectionate communication accelerates neuroendocrine stress recovery. Health Commun. 2007;22(2):123-32. doi: 10.1080/10410230701454015. PMID 17668992